CLINICAL TRIAL: NCT04224246
Title: Impact of Gamma-OH on Sleep in ICU Patients Difficult to Wean from Mechanical Ventilation
Brief Title: Impact of Gamma-OH on Sleep in ICU Patients
Acronym: GO-SLEEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-SLEEP
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Weaning from Mechanical Ventilation
MeSH Terms: interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One arm with Gamma-OH® treatment (Experimental): Gamma-OH® will be administered intravenously at a dose of 20 mg/kg/h for 6 hours between 10 p.m. to 4 a.m.
  Interventions: Drug: Gamma Hydroxybutyrate

INTERVENTIONS:
Drug: Gamma Hydroxybutyrate — Gamma-OH® will be administered intravenously at a dose of 20 mg/kg/h for 6 hours

SUMMARY:
The Main objective of the trial is to assess sleep quality with Gamma-OH® in patients difficult to wean from mechanical ventilation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* intubated at least 24 hours
* difficult weaning from mechanical ventilation according to international guidelines, i.e. who failed at least one spontaneous breathing trial.
* Patients will be included after to obtain inform consent.

Exclusion Criteria:

* neuromuscular disease
* central nervous disease
* psychiatric disease
* severe obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having poor sleep with Gamma-OH | Hour24
  Primary end point will be analyzed from sleep recordings performed during a single night with Gamma-OH®.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, Poitiers, France